CLINICAL TRIAL: NCT04241341
Title: A Randomized Controlled Trial: Does Immediate Lymphatic Reconstruction Decrease the Incidence of Lymphedema After Axillary Lymph Node Dissection
Brief Title: Does Immediate Lymphatic Reconstruction Decrease the Risk of Lymphedema After Axillary Lymph Node Dissection
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-021
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Lymphedema
Keywords: Axillary Lymph Node Dissection; Lymphatic Reconstruction; 20-021
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two groups:
  ALND with ILR (intervention group) and ALND without ILR (control group; current standard treatment at Memorial Sloan Kettering [MSK]).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- axillary lymph node dissection with ILR (Experimental)
  Interventions: Procedure: Axillary Lymph Node Dissection with Immediate Lymphatic Reconstruction; Other: quality-of-life questionnaires; Other: measured by arm volume
- axillary lymph node dissection (ALND) without ILR (Active Comparator)
  Interventions: Procedure: Axillary Lymph Node Dissection without Immediate Lymphatic Reconstruction; Other: quality-of-life questionnaires; Other: measured by arm volume

INTERVENTIONS:
Procedure: Axillary Lymph Node Dissection with Immediate Lymphatic Reconstruction — Axillary Lymph Node Dissection with Immediate Lymphatic Reconstruction
  Arms: axillary lymph node dissection with ILR
Procedure: Axillary Lymph Node Dissection without Immediate Lymphatic Reconstruction — Current standard treatment at Memorial Sloan Kettering [MSK]).
  Arms: axillary lymph node dissection (ALND) without ILR
Other: quality-of-life questionnaires — Four validated patient reported outcome measures (PROMs): the Upper Limb Lymphedema-27 (ULL-27), the Quality of Life Measure for Limb Lymphedema (LYMQOL), the Center for Epidemiologic Studies Depression Scale-Revised (CESD-R), and the Beck Anxiety Inventory (BAI). Study participants will undergo standard lymphedema measurements and quality-of-life questionnaires at baseline before ALND and postoperatively at 6 weeks (+/- 30 days) and at 6, 12, 18, and 24 months (+/- 30 days). If patients are unable to complete their questionnaires at the time of their in-office visit, a link to the questionnaires in REDCap will be emailed to them.
Other: measured by arm volume — Bilateral arm volumes will be measured with sequential circumferential measurements with the truncated cone formula. If a patient cannot return to Manhattan for these assessments but is seen by a lymphedema therapist in a regional location or at an institution outside of MSK as part of their routine cancer treatment, this data can be used in the final analysis

SUMMARY:
The researchers are doing this study to see if having immediate lymphatic reconstruction after axillary lymph node dissection (ALND) can decrease the development of lymphedema, a side effect of ALND. Other purposes of the study include:

Comparing the approach of immediate lymphatic reconstruction after ALND with the approach of ALND alone Looking at whether having immediate lymphatic reconstruction after ALND improves a person's quality of life Seeing if adding standard of care radiation therapy to either study approach (immediate lymphatic reconstruction after ALND or ALND alone) has an effect on development of lymphedema

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients 18-75 years of age
* Patients consenting for unilateral ALND (prior history of SLNBx allowed if <6 months from consent) OR patients consenting for unilateral SLNBx with possible ALND, with a clinically or radiographically positive lymph node OR a high likelihood of ALND per the Breast Surgeon
* Identification of at least one transected lymphatic channel and at least one vein to be used for bypass at the time of ALND during surgery

Exclusion Criteria:

* Male breast cancer patients
* Non-English speaking participants
* Female breast cancer patients with axillary recurrence
* Female breast cancer patients who have a history of ALND
* Female patients requiring bilateral ALND for the treatment of their breast cancer
* Female breast patients treated with SLNBx only

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 180 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
the number of patients that had a decrease incidence of lymphedema | up to 2 years
  as measured by arm volume will be a ≥10% increase in arm volume

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Coriddi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent and Followup), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm